CLINICAL TRIAL: NCT06688487
Title: Early Postoperative Extubation in Hypoxemic ICU Patients: a Multicenter, Randomized Controlled Trial
Brief Title: Postoperative Extubation in Hypoxemic Patients
Acronym: EPHYRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00535-42
Record Dates: First submitted 2024-10-17; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hypoxemia; Extubation; Postoperative Respiratory Complication
Keywords: extubation; hypoxemia; postoperative respiratory complication; weaning; facilitative non invasive strategy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypoxemic extubation group (Experimental): Randomized patients exhibit relative hypoxemia, defined by an SpO2 ≤ 90% while receiving 6 liters of oxygen or FiO2 of 40%. They must not have severe hypoxemia, defined as an SpO2 < 86% while receiving 9 liters of oxygen or FiO2 of 50%. Additionally, they must not show clinical signs of poor tolerance to the spontaneous breathing trial. Patients randomized to the "hypoxemic extubation group" are extubated despite the presence of relative hypoxemia after one hour of reventilation. Following extubation, a non-invasive oxygenation strategy is initiated, alternating between non-invasive ventilation and high-flow oxygen therapy for a minimum of 24 hours.
  Interventions: Other: early extubation of hypoxemic patients
- conventional extubation group (No Intervention): Patients in the conventional extubation group also present with relative hypoxemia, defined as an SpO2 ≤ 90% on 6 liters of oxygen or FiO2 of 40% at the time of randomization, but they will only be extubated after correction of this hypoxemia. In practice, patients in the conventional extubation group are not extubated after randomization and continue on invasive ventilation. A new spontaneous breathing trial (SBT) can be performed between 2 and 6 hours after randomization, and if unsuccessful, it may be repeated daily at the discretion of the clinician. Patients in the conventional extubation group will only be extubated when their SpO2 exceeds 90% during an SBT conducted on 6 liters of oxygen or FiO2 of 40%.
  After extubation, a non-invasive oxygenation strategy will be initiated, alternating between non-invasive ventilation (NIV) and high-flow oxygen therapy, for a minimum of 24 hours.

INTERVENTIONS:
Other: early extubation of hypoxemic patients — patient extubated after the spontaneous ventilation trial despite the presence of hypoxemia defined by SpO2 ≤ 90% either in T-piece under 6 L/min, or under FiO2 = 40% if SBT is performed in spontaneous ventilation with minimal inspiratory assistance.
  Arms: hypoxemic extubation group

SUMMARY:
The objective of this clinical trial is to assess whether early extubation of patients with hypoxemia during the spontaneous breathing trial (SBT) shortens the duration of ventilatory support. The trial will also evaluate the safety of this approach. The key research questions include:

Does early extubation of hypoxemic patients reduce the total duration of ventilatory support (both invasive and non-invasive) by 36 hours? Does early extubation of hypoxemic patients increase the number of ventilator-free days by day 28? Can the safety of early extubation in hypoxemic patients be ensured by confirming no significant differences in rates of reintubation, tracheostomy, or mortality? The trial will compare ventilatory outcomes between two groups: hypoxemic patients who undergo early extubation (hypoxemic extubation group) and those who remain on invasive ventilation until hypoxemia resolves (conventional extubation group).

DETAILED DESCRIPTION:
International guidelines recommend extubating patients after correction of hypoxemia, meaning if the SpO2 measured during the spontaneous breathing trial is above 92%. However, there is strong rationale for modifying this practice to extubate patients earlier, particularly those presenting with hypoxemia after major surgery, by using alternating non-invasive ventilation (NIV) and high-flow oxygen therapy:

Several studies have found no link between patient oxygenation and extubation success, where outcomes for hypoxemic and non-hypoxemic patients are similar. Isolated hypoxemia thus does not appear to be a predictor of reintubation.

Hypoxemia is very common following major surgery, primarily due to shunts caused by atelectasis. Treatment for these atelectasis includes airway pressurization, bronchial secretion drainage, mobilization, and reducing factors that lead to diaphragmatic dysfunction.

In patients on invasive mechanical ventilation, secretion drainage is impaired, and mobilization to a seated position is more challenging. It has also been shown that diaphragmatic dysfunction occurs with prolonged ventilation. Hypoxemia can therefore be sustained by invasive ventilation, increasing the risk of therapeutic escalation.

Current guidelines do not account for the widespread use of non-invasive assistance techniques (such as high-flow oxygen therapy and non-invasive ventilation) that are now routinely employed in intensive care. These techniques allow for adequate oxygenation with high patient comfort and good tolerance.

Prolonging invasive ventilation in hypoxemic patients, as recommended by guidelines, could lead to associated complications. In contrast, early extubation of patients with hypoxemia may reduce the duration of both invasive and non-invasive ventilation, as well as complications related to prolonged invasive ventilation, without increasing the risk of reintubation.

Compared to continuing mechanical ventilation until hypoxemia is corrected, extubating purely hypoxemic patients and transitioning them to non-invasive ventilation techniques could represent a significant improvement in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Francophone patient affiliated to a health insurance plan;
* Patient having granted free, informed and written consent to participate in the study;
* Patient with hypoxemia defined as SpO2 ≤ 90% under 6 L/min or FiO2 40% during spontaneous breathing trial.

Exclusion Criteria:

* Presence of hypercapnia at the end of SBT (PaCO2 above 50 mmHg);
* Presence of severe hypoxemia during SBT defined by SpO2 below 86% under 9 L/min or FiO2 = 50%;
* Presence of poor clinical tolerance of SBT defined by polypnoea above 30/min, agitation, sweating, hypertension (PAS above 180 mmHg), tachycardia (HR above 140 bpm) or arrhythmia;
* Presence of an ineffective cough or major bronchial congestion;
* Patient already included in a type 1 interventional research protocol (RIPH1), modifying the procedure for ventilatory weaning and/or ventilatory support after extubation;
* Anatomical factors precluding the use of NIV or high-flow oxygen therapy, notably facial or cervico-facial malformations;
* Tracheostomized patient;
* History of obstructive ventilatory disorders with indication for NIV post-extubation, chronic obstructive pulmonary disease (COPD) GOLD score III/IV;
* History of obstructive sleep apnea syndrome with equipment;
* cardiogenic pulmonary edema;
* Patient on extracorporeal membrane oxygenation (ECMO) at the time of inclusion;
* Patient under guardianship or curatorship;
* Minor patients;
* Patient deprived of liberty or under court protection;
* Pregnant or breast-feeding women;
* Patient in therapeutic limitation with decision not to re-intubate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
time to ventilatory weaning | from date of randomisation until the date of cessation of non invasive ventilation or death from any cause, assessed up to 90 days after randomization
  Time in hours from randomization to discontinuation of ventilatory support (invasive and non-invasive).

SECONDARY OUTCOMES:
neuromyopathie score | day 7of randomisation/day of weaning from non-invasive ventilation
  MRC score assessed in each group on day 7 of randomisation and on the day of weaning from non-invasive ventilation.
death | at 28 and 90 days after randomisation
  occuring of death during ICU, hospital management and at day 90
ventilatory support duration between randomization and day 28 | from randomisation to day 28
  Number of days alive without ventilation (invasive or non-invasive) at day 28 of randomization.
invasive ventilation duration | from date of randomisation until the date of cessation of invasive ventilation or death from any cause whichever came first assessed up to 90 days after randomization
  Time in hours between randomization and cessation of invasive ventilation
non invasive ventilation duration | from date of extubation until the date of cessation of non invasive ventilation strategy or date of reintubation assessed up to 90 days
  Time in hours between initiation and cessation of non-invasive support after extubation
reintubation rate | up to day 90 after randomisation
  Number of patients requiring reintubation
Rate of ventilator-associated pneumonia. | up to day 90 after randomisation
  Episodes of ventilator-associated pneumonia according to specific definition
Rate of pneumonia not acquired under invasive mechanical ventilation | up to 90 days after randomisation
  Epiodes of pneumonia not acquired during invasive mechanical ventilation
time to mobilisation | from date of randomisation until the date of the first chair mobilization or death from any cause whichever came first , assessed up to 90 days after randomization
  time in hours between randomization and the first mobilisation in the chair
time to ambulation | from date of randomisation until the date of the first ambulation or death from any cause whichever came first , assessed up to 90 days after randomization
  time in hours between randomization and first ambulation
length of stay in ICU | from date of entrance until the date of discharge to ICU or death from any cause whichever came first assessed up to 52 weeks after randomization
  number of day between admission and discharge to ICU
length of stay in ICU after randomisation | from randomisation until the date of discharge to ICU or death from any cause whichever came first assessed up to 52 weeks after randomization
  number of day between randomisation and discharge from the ICU
length of stay in hospital after randomisation | from date of randomisation until the date of hospital discharge or death from any cause whichever came first assessed up to 52 weeks after randomization
  Time in days from randomisation to hospital discharge
length of stay in hospital | from date of admission until the date of hospital discharge or death from any cause whichever came first assessed up to 52 weeks after randomization
  number of day between admission to discharge of hospital

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - centre hospitalier Victor Dupouy, Argenteuil
  - CHRU de Besançon, Besançon
  - Marie Lannelongue Hospital, Le Plessis-Robinson
  - Hôpital Saint Eloi, CHU Montpellier, Montpellier
  - CHU la pitié salpêtrière, Paris
  - CHU la pitié Salpêtrière, Paris
  - Institut mutualiste Montsouris, Paris
  - réanimation polyvalente hopital saint joseph groupe hospitalier Paris saint Joseph, Paris
  - hôpital george Pompidou, Paris
  - CHU de Reims, Reims
  - Centre Cardiologique Du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Background] Quintard H, l'Her E, Pottecher J, Adnet F, Constantin JM, De Jong A, Diemunsch P, Fesseau R, Freynet A, Girault C, Guitton C, Hamonic Y, Maury E, Mekontso-Dessap A, Michel F, Nolent P, Perbet S, Prat G, Roquilly A, Tazarourte K, Terzi N, Thille AW, Alves M, Gayat E, Donetti L. Experts' guidelines of intubation and extubation of the ICU patient of French Society of Anaesthesia and Intensive Care Medicine (SFAR) and French-speaking Intensive Care Society (SRLF) : In collaboration with the pediatric Association of French-speaking Anaesthetists and Intensivists (ADARPEF), French-speaking Group of Intensive Care and Paediatric emergencies (GFRUP) and Intensive Care physiotherapy society (SKR). Ann Intensive Care. 2019 Jan 22;9(1):13. doi: 10.1186/s13613-019-0483-1. PMID 30671726
- [Background] Perkins GD, Mistry D, Gates S, Gao F, Snelson C, Hart N, Camporota L, Varley J, Carle C, Paramasivam E, Hoddell B, McAuley DF, Walsh TS, Blackwood B, Rose L, Lamb SE, Petrou S, Young D, Lall R; Breathe Collaborators. Effect of Protocolized Weaning With Early Extubation to Noninvasive Ventilation vs Invasive Weaning on Time to Liberation From Mechanical Ventilation Among Patients With Respiratory Failure: The Breathe Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1881-1888. doi: 10.1001/jama.2018.13763. PMID 30347090